CLINICAL TRIAL: NCT02145286
Title: A Phase I/II Single Arm Prospective Single Fraction Real-time Stereotactic Body Radiation Therapy Dose Escalation Trial of Rapid Helical TomoTherapy-based Radiation Therapy for Patients With Painful Osseous Metastatic Disease
Brief Title: Phase 1/2 Study to Determine Optimal Dose for Treating Bone Metastases Using Novel STAT-RT Workflow
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Paul W. Read, MD (Other)
Responsible Party: Sponsor-Investigator, Paul W. Read, MD, Professor, University of Virginia
Organization: University of Virginia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16964
Record Dates: First submitted 2014-05-19; First posted 2014-05-22 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Metastatic Bone Lesion
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiation Therapy (Experimental): Stereotactic Body Radiation Therapy
  Interventions: Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy — SBRT is a high dose and highly conformal radiation dose treatment with the goal of rapid tumor killing and/or ablation of tumors

SUMMARY:
The purpose of this research study is to evaluate the safety and effectiveness of an experimental procedure called Focused Radiation that may result in a faster way to plan and deliver radiation for the treatment of pain caused by metastatic bone tumors (cancerous tumors that originally came from another organ and have spread to bones). In this trial a single fraction of radiation will be given from 8-15 Gray.

DETAILED DESCRIPTION:
The purpose of this research study is to evaluate the safety and effectiveness of an experimental procedure called Focused Radiation that may result in a faster way to plan and deliver radiation for the treatment of pain caused by metastatic bone tumors (cancerous tumors that originally came from another organ and have spread to bones).

Focused radiation (the radiation is focused on the tumor in the bone with reduced radiation dose to the normal tissues) is used as standard of care treatment for patients with painful metastatic tumors in their spines with just one treatment. In this study, the focused radiation will be used to treat tumors in other bones as well. The current standard of care radiation treatment planning and delivery can take 2 to 3 weeks from start to finish depending on how many treatments are given although the standard of care is to treat patients with 1-10 treatments. The University of Virginia has developed an experimental workflow/process: a radiation treatment planning and delivery workflow called "STAT RAD" (STAT means "right away", and RAD means radiation). This experimental workflow will shorten the time it takes to plan and treat painful bone metastases to 1-2 hours.

When only one treatment is given the standard radiation dose is 8 Gray. This has resulted in radiation retreatment rates to the treated bone of 20% in prior studies for persistent or recurrent bone pain. In this study patients will be treated with higher doses of targeted radiation to determine if higher doses, which have been reported to be safely delivered for bone metastases in the spine with very low re-treatment rates, can be safely delivered to non-spine bone metastases. After the treatment, patients will be followed for pain relief in the treated bone, need for pain medication, quality of life, toxicity, and the need to retreat the bone metastasis for persistent or recurrent pain.

ELIGIBILITY:
Inclusion Criteria:

* Patient has 1-3 major painful osseous metastases (target lesions)
* Radiographic evidence (CT, MR, or PET CT) consistent with osseous metastatic disease on CT, MR, or PET CT obtained within 4 weeks of treatment will be used for pre-study treatment delivery. The GTV of the target lesions will be determined from this radiographic study and must be ≤ 250 cubic centimeters.

NOTE: Patient is still eligible if a diagnostic image set is not available within 4 weeks of treatment if the patient will undergo a kVCT simulation in the Department of Radiation Oncology with contouring directly onto this image set.

* Patient is medically able to undergo palliative radiation therapy
* Patient has pain that is persistent and distinguishably associated with the target sites to be treated
* Planning Target Volume 1 (PTV1) must be > 5mm from the spinal cord or brain
* Women of Childbearing age and men must consent to use adequate contraception for six months following study entry

Exclusion Criteria:

* Inability to lie on the treatment table for 1 hour
* Systemic therapeutic radionuclide delivery within 30 days prior to treatment
* Target lesions have been previously treated with external beam radiation
* Long bone target lesions with a Mirels fracture score >7
* Unstable bone in the target lesion requiring surgical stabilization
* PTV1 is located within 5mm of spinal cord or brain
* A serious, uncontrolled medical disorder
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2013-10; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Radiation Dose | Up to 12 months following treatment
  Determine the optimal dose range for treatment of osseous bone metastases with single SBRT (Stereotactic Body Radiation Therapy) treatment using the STAT RAD (right away/radiation) workflow

SECONDARY OUTCOMES:
Single Treatment Pain Scores | Up to 4 weeks following treatment
  Patients will complete questionnaires to determine whether the treatment of osseous bone metastases with single treatment using the STAT RAD workflow results in a significant change in pain scores at 4 weeks following treatment of patients with good prognosis, compared to baseline scores
Paired Dose Pain Score Comparison | Up to 4 weeks following treatment
  Patient questionnaires will be used to estimate the difference in the mean change in pain score from baseline to 4 weeks following treatment of patients with good prognosis between pairs of dose levels among those in the range of optimal doses
Post Treatment Measures | Up to 12 months following treatment
  Patients will complete questionnaires to capture pain scores of the treated lesion(s), analgesic use, patient functional status, patient quality of life, and patient satisfaction at 1,4,8, and 12 weeks and at 6 and 12 months following treatment. Rates of radiation-retreatment within one year will also be captured for the treated target lesion(s).

CONTACTS AND LOCATIONS:
Overall Officials: Paul W Read, MD, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No